CLINICAL TRIAL: NCT03171038
Title: Long-term Impact of a 6-months Telemedical Care Program on Mortality, Readmissions and Healthcare Costs in Patients With Chronic Heart Failure The TElemonitoring in the Management of Heart Failure (TEMA-HF) 1 Long-term Follow-up Study
Brief Title: The TElemonitoring in the Management of Heart Failure (TEMA-HF) 1 Long-term Follow-up Study
Acronym: TEMA-HFLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, Prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jessa Hospital
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Telemonitoring in Coronary Artery Disease
Keywords: Telemonitoring; Chronic Heart Failure; eHealth; Mortality

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring group (Experimental): 6 months of telemonitoring (t0-t1), followed by usual care up until common long-term stopping date (t1-t2).
  Interventions: Other: Telemonitoring
- Usual care group (No Intervention): Usual care from t0 up until the common stopping date (t2).

INTERVENTIONS:
Other: Telemonitoring
  Arms: Telemonitoring group

SUMMARY:
TEMA-HF 1 Long-Term Follow-up study is a follow-up study of TEMA-HF 1. It assessed the long-term impact of a 6-months telemonitoring program in chronic heart failure patients.

DETAILED DESCRIPTION:
The telemonitoring (TM) group patients received a 6-months TM program, followed by standard heart failure care until the long-term follow-up evaluation.

The usual care (UC) patients received ususal care during the first six months, followed by standard heart failure care until the long-term follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure patients
* Treated for heart failure according to current guidelines
* ≥ 18 years of age
* Able to provide informed consent

Exclusion Criteria:

* Reversible forms of acute heart failure (myocarditis)
* Presence of severe aortic stenosis
* Previous residency in a nursing home
* Inclusion in a cardiac rehabilitation program on discharge
* Chronic kidney disease stage ≥ 4
* Planned dialysis in the next six months
* Life expectancy < 1 year due to non-heart failure related reasons
* Severe chronic obstructive pulmonary disease, GOLD ≥ III
* Cognitive and/or mental problems interfering with the performance of daily measurements and data transmission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2015-08-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Start of study to long-term follow-up (6.5 years).
  All-cause mortality

SECONDARY OUTCOMES:
days lost due to heart failure readmissions | Start of study to long-term follow-up (6.5 years).
  days lost due to heart failure readmissions
days lost due to all readmissions | Start of study to long-term follow-up (6.5 years).
  days lost due to all readmissions
days lost due to death or heart failure readmissions | Start of study to long-term follow-up (6.5 years).
  days lost due to death or heart failure readmissions
percentage of follow-up time spent in hospital for heart failure | Start of study to long-term follow-up (6.5 years).
  percentage of follow-up time spent in hospital for heart failure
percentage of follow-up time spent in hospital for all reasons | Start of study to long-term follow-up (6.5 years).
  percentage of follow-up time spent in hospital for all reasons
percentage of follow-up time lost to death or heart failure readmissions | Start of study to long-term follow-up (6.5 years).
  percentage of follow-up time lost to death or heart failure readmissions

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frederix I, Vanderlinden L, Verboven AS, Welten M, Wouters D, De Keulenaer G, Ector B, Elegeert I, Troisfontaines P, Weytjens C, Mullens W, Dendale P. Long-term impact of a six-month telemedical care programme on mortality, heart failure readmissions and healthcare costs in patients with chronic heart failure. J Telemed Telecare. 2019 Jun;25(5):286-293. doi: 10.1177/1357633X18774632. Epub 2018 May 10. PMID 29742959